CLINICAL TRIAL: NCT03859804
Title: Comparison of Pain Levels in Fusion Prostate Biopsy and Standard TRUS-Guided Biopsy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: TC Erciyes University (Other)
Responsible Party: Principal Investigator, Abdullah Demirtas, Abdullah Demirtas, Md, Assoc. Prof., TC Erciyes University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 2014/508
Record Dates: First submitted 2019-02-24; First posted 2019-03-01 (Actual); Last update posted 2019-03-01 (Actual); Status verified 2019-02

CONDITIONS: Pain Due to Certain Specified Procedures; Prostate Cancer; Biopsy
Keywords: fusion; prostate; biopsy; pain
MeSH Terms: conditions — Prostatic Neoplasms; Pain

STUDY DESIGN:
Intervention Model Description: pain levels after standard transrectal prostate 12 core biopsy and MRI -US fusion prostate biopsy were detected and compared in 2 groups.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group 1 (Experimental): In Group 1, Patients detected with a PI-RADS (Prostate Imaging Reporting and Data System) ≥3 lesion on MpMRI underwent MpMRI-guided MRI- US fusion prostate biopsy. In this fusion biopsy, 12 core standard biopsy and 2-4 cores of biopsies from lesions defined on multiparametric prostate MRI
  Interventions: Procedure: MRI- US fusion prostate biopsy (FPB)
- Group 2 (Active Comparator): In Group 2, patients who had no suspected lesions or had a PI-RADS <3 lesion on MpMRI underwent Transrectal ultrasound guided 12 core prostate biopsy (SPB).
  Interventions: Procedure: Standard transrectal 12 core biopsy

INTERVENTIONS:
Procedure: Standard transrectal 12 core biopsy — TRUS-guided SPB was performed by obtaining 12 core samples in each patient. 6 cores from left and right. the cores labeled as, apex, mid, base, apex far lateral, mid far lateral and base far lateral
  Other Names: Group 2
  Arms: Group 2
Procedure: MRI- US fusion prostate biopsy (FPB) — FPB was performed by obtaining 10-12 core samples in each patient, followed by the acquisition of 2-4 core samples for each suspected lesion detected on MpMRI (combined biopsy)
  Other Names: Group 1
  Arms: Group 1

SUMMARY:
The aim of this study was to compare the pain levels in transrectal ultrasound (TRUS)-guided standard 12-core prostate biopsy (SPB) and multiparametric prostate magnetic resonance imaging (MpMRI)-guided fusion prostate biopsy (FPB).

DETAILED DESCRIPTION:
The study included patients that underwent prostate biopsy under local anesthesia (intrarectal 2% lidocaine gel + periprostatic nerve block) due to suspected prostate cancer. Patients detected with a Prostate Imaging Reporting and Data System score (PIRADS) ≥3 lesion on MpMRI underwent MpMRI-guided FPB (Group I) and the patients who had no suspected lesions or had a PI-RADS <3 lesion on MpMRI underwent TRUS-guided SPB (Group II). Pain assessment was performed using Visual Analog Scale (VAS) 5 min after the procedure. Following the procedure, the patients were asked to indicate the most painful biopsy step among the three steps (1: insertion of the probe into the rectum, 2: probe manipulation, 3: the piercing of the biopsy needle).

ELIGIBILITY:
Inclusion Criteria:

* Elevated blood prostate specific antigen (PSA) levels according to patients age. PSA >2ng/ml for whom aged between 50-60, and PSA >4ng/ml for whom were above 60 years old
* Having suspicious digital rectal examination
* having multi-parametric prostate MRI before prostate biopsy
* Having MRI defined lesions which were PIRADS - 3 -4-5

Exclusion Criteria:

* PSA > 50 ng/ml
* previous negative biopsy
* neurological disorders that could affect the pain level such as paraplegia or hemiplegia, analgesics use for any reason on the day of or the day before the procedure,
* patients underwent biopsy under general anesthesia,
* having such diseases as anal fissure or hemorrhoidal disease that could alter the pain threshold

Ages: 50 Years to 75 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 252 (Actual)
Dates: Start 2016-12-01 (Actual); Primary Completion 2019-01-31 (Actual); Study Completion 2019-02-01 (Actual)

PRIMARY OUTCOMES:
To detect painful steps of biopsy procedure by asking patients verbally | Within 5 minutes after biopsy
  to ask patients most painful step of procedure that verbally defined them before biopsy as 1: insertion of the probe into the rectum, 2: probe manipulation, and 3: the piercing of the biopsy needle
Over all Visual analogue Score (VAS) score of procedure(From 0 to 100 points, 100 is max pain score according to patient) | Within 5 minutes after prostate biopsy
  pain assessment was performed using Visual Analogue Scale (VAS)

CONTACTS AND LOCATIONS:
Overall Officials: Abdullah T Demirtaş, MD, Principal Investigator — Erciyes University Faculty of Medicine Department of Urolgoy
Locations (1):
- Department of Urology, Ercieys University, Faculty Of Medicine,, Kayseri, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Ferlay J, Soerjomataram I, Dikshit R, Eser S, Mathers C, Rebelo M, Parkin DM, Forman D, Bray F. Cancer incidence and mortality worldwide: sources, methods and major patterns in GLOBOCAN 2012. Int J Cancer. 2015 Mar 1;136(5):E359-86. doi: 10.1002/ijc.29210. Epub 2014 Oct 9. PMID 25220842
- [Background] Siddiqui MM, Rais-Bahrami S, Turkbey B, George AK, Rothwax J, Shakir N, Okoro C, Raskolnikov D, Parnes HL, Linehan WM, Merino MJ, Simon RM, Choyke PL, Wood BJ, Pinto PA. Comparison of MR/ultrasound fusion-guided biopsy with ultrasound-guided biopsy for the diagnosis of prostate cancer. JAMA. 2015 Jan 27;313(4):390-7. doi: 10.1001/jama.2014.17942. PMID 25626035
- [Background] Gayet M, van der Aa A, Beerlage HP, Schrier BP, Mulders PF, Wijkstra H. The value of magnetic resonance imaging and ultrasonography (MRI/US)-fusion biopsy platforms in prostate cancer detection: a systematic review. BJU Int. 2016 Mar;117(3):392-400. doi: 10.1111/bju.13247. Epub 2015 Aug 28. PMID 26237632
- [Background] Hwang SI, Lee HJ, Lee SE, Hong SK, Byun SS, Lee SC, Choe G. Value of MR-US fusion in guidance of repeated prostate biopsy in men with PSA < 10 ng/mL. Clin Imaging. 2019 Jan-Feb;53:1-5. doi: 10.1016/j.clinimag.2018.09.012. Epub 2018 Sep 22. PMID 30265884
- [Background] Mannaerts CK, Kajtazovic A, Lodeizen OAP, Gayet M, Engelbrecht MRW, Jager GJ, Wijkstra H, de Reijke TM, Beerlage HP. The added value of systematic biopsy in men with suspicion of prostate cancer undergoing multiparametric MRI-targeted biopsy. Urol Oncol. 2019 May;37(5):298.e1-298.e9. doi: 10.1016/j.urolonc.2019.01.005. Epub 2019 Jan 17. PMID 30660493
- [Background] Luan Y, Huang TB, Gu X, Zhou GC, Lu SM, Tao HZ, Liu BD, Ding XF. Effect of prostate volume on the peripheral nerve block anesthesia in the prostate biopsy: A strobe-compliant study. Medicine (Baltimore). 2016 Jul;95(28):e4184. doi: 10.1097/MD.0000000000004184. PMID 27428215
- [Background] Fourcade A, Payrard C, Tissot V, Perrouin-Verbe MA, Demany N, Serey-Effeil S, Callerot P, Coquet JB, Doucet L, Deruelle C, Joulin V, Nonent M, Fournier G, Valeri A. The combination of targeted and systematic prostate biopsies is the best protocol for the detection of clinically significant prostate cancer. Scand J Urol. 2018 Jun;52(3):174-179. doi: 10.1080/21681805.2018.1438509. Epub 2018 Feb 20. PMID 29463177
- [Result] Autorino R, De Sio M, Di Lorenzo G, Damiano R, Perdona S, Cindolo L, D'Armiento M. How to decrease pain during transrectal ultrasound guided prostate biopsy: a look at the literature. J Urol. 2005 Dec;174(6):2091-7. doi: 10.1097/01.ju.0000181212.51025.06. PMID 16280735
- [Result] Mazdak H, Abtahi AM, Momeni F, Izadpanahi MH. A comparison of pain control and complications using three different ways of anesthesia in patients undergoing transrectal ultrasound-guided prostate biopsy. J Res Med Sci. 2018 Feb 20;23:17. doi: 10.4103/jrms.JRMS_639_17. eCollection 2018. PMID 29531569
- [Result] Wang N, Fu Y, Ma H, Wang J, Gao Y. Advantages of caudal block over intrarectal local anesthesia plus periprostatic nerve block for transrectal ultrasound guided prostate biopsy. Pak J Med Sci. 2016 Jul-Aug;32(4):978-82. doi: 10.12669/pjms.324.9823. PMID 27648052
- [Result] Yang Y, Liu Z, Wei Q, Cao D, Yang L, Zhu Y, Wei X, Tang Z, Liu L, Han P. The Efficiency and Safety of Intrarectal Topical Anesthesia for Transrectal Ultrasound-Guided Prostate Biopsy: A Systematic Review and Meta-Analysis. Urol Int. 2017;99(4):373-383. doi: 10.1159/000481830. Epub 2017 Oct 30. PMID 29084411
- [Result] Alabi TO, Tijani KH, Adeyomoye AA, Jeje EA, Anunobi CC, Ogunjimi MA, Ojewola RW, Akanmu ON, Oliyide AE, Orakwe DE. Combined intrarectal lidocaine gel and periprostatic nerve block: A 'balanced' anaesthesia for transrectal ultrasound-guided prostate biopsy? Niger Postgrad Med J. 2018 Oct-Dec;25(4):252-256. doi: 10.4103/npmj.npmj_145_18. PMID 30588947
- [Result] Collins GN, Lloyd SN, Hehir M, McKelvie GB. Multiple transrectal ultrasound-guided prostatic biopsies--true morbidity and patient acceptance. Br J Urol. 1993 Apr;71(4):460-3. doi: 10.1111/j.1464-410x.1993.tb15993.x. PMID 8499991
- [Result] Hollingsworth JM, Miller DC, Wei JT. Local anesthesia in transrectal prostate biopsy. Urology. 2006 Jun;67(6):1283-4. doi: 10.1016/j.urology.2005.12.016. PMID 16765193
- [Result] Robins D, Lipsky M, RoyChoudry A, Wenske S. Assessment of Discomfort and Pain in Patients Undergoing Fusion Magnetic Resonance Imaging-guided vs TRUS-guided Prostate Biopsy. Urology. 2018 Jun;116:30-34. doi: 10.1016/j.urology.2018.02.029. Epub 2018 Mar 12. PMID 29545039
- [Result] Arsov C, Rabenalt R, Quentin M, Hiester A, Blondin D, Albers P, Antoch G, Schimmoller L. Comparison of patient comfort between MR-guided in-bore and MRI/ultrasound fusion-guided prostate biopsies within a prospective randomized trial. World J Urol. 2016 Feb;34(2):215-20. doi: 10.1007/s00345-015-1612-6. Epub 2015 Jun 9. PMID 26055645
- [Result] Fabiani A, Servi L, Filosa A, Fioretti F, Maurelli V, Tombolini F, Talle M, Mammana G. May ultrasound probe size influence pain perception of needle piercing during transrectal prostate biopsy? A prospective evaluation. Arch Ital Urol Androl. 2016 Oct 5;88(3):223-227. doi: 10.4081/aiua.2016.3.223. PMID 27711100
- [Result] Yan P, Wang XY, Huang W, Zhang Y. Local anesthesia for pain control during transrectal ultrasound-guided prostate biopsy: a systematic review and meta-analysis. J Pain Res. 2016 Oct 11;9:787-796. doi: 10.2147/JPR.S117451. eCollection 2016. PMID 27785093
- [Result] Urabe F, Kimura T, Shimomura T, Onuma H, Yamamoto T, Sasaki H, Miki J, Kuruma H, Miki K, Egawa S. Prospective comparison of the efficacy of caudal versus periprostatic nerve block, both with intrarectal local anesthesia, during transrectal ultrasonography-guided prostatic needle biopsy. Scand J Urol. 2017 Aug;51(4):245-250. doi: 10.1080/21681805.2017.1318299. Epub 2017 Apr 26. PMID 28443752
- [Result] Valdez-Flores RA, Campos-Salcedo JG, Torres-Gomez JJ, Sedano-Lozano A, Pares-Hipolito J, Shelton LM, Canizalez-Roman A, Valdez-Flores MA. Prospective comparison among three intrarectal anesthetic treatments combined with periprostatic nerve block during transrectal ultrasonography-guided prostate biopsy. World J Urol. 2018 Feb;36(2):193-199. doi: 10.1007/s00345-017-2136-z. Epub 2017 Nov 23. PMID 29170792
- [Result] Gomez-Gomez E, Ramirez M, Gomez-Ferrer A, Rubio-Briones J, Iborra I, J Carrasco-Valiente, Campos JP, Ruiz-Garcia J, Requena-Tapia MJ, Solsona E. Assessment and clinical factors associated with pain in patients undergoing transrectal prostate biopsy. Actas Urol Esp. 2015 Sep;39(7):414-9. doi: 10.1016/j.acuro.2015.01.007. Epub 2015 Mar 6. English, Spanish. PMID 25745791
- [Result] Bastide C, Lechevallier E, Eghazarian C, Ortega JC, Coulange C. Tolerance of pain during transrectal ultrasound-guided biopsy of the prostate: risk factors. Prostate Cancer Prostatic Dis. 2003;6(3):239-41. doi: 10.1038/sj.pcan.4500664. PMID 12970728
- [Result] Djavan B, Waldert M, Zlotta A, Dobronski P, Seitz C, Remzi M, Borkowski A, Schulman C, Marberger M. Safety and morbidity of first and repeat transrectal ultrasound guided prostate needle biopsies: results of a prospective European prostate cancer detection study. J Urol. 2001 Sep;166(3):856-60. PMID 11490233